CLINICAL TRIAL: NCT04982861
Title: Bioequivalence Study of Cefixime Trihydrate 100 mg/5 mL DS in Indonesia Healthy Volunteers
Brief Title: Bioequivalence Study of Cefixime Trihydrate Dry Syrup in Indonesia Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PT Bernofarm (Industry)
Collaborators: PT Pharma Metric Labs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 432/STD/PML/2018
Record Dates: First submitted 2021-07-23; First posted 2021-07-29 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Drug Use
Keywords: bioequivalence study; cefixime trihydrate; dry syrup; Indonesia
MeSH Terms: interventions — Cefixime; Suspensions

STUDY DESIGN:
Intervention Model Description: Randomized, single-blind, two-period, single dose, cross-over design in 22 healthy subjects under fasting condition.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cefixime trihydrate 100 mg/5 mL dry syrup (Experimental): Cefixime trihydrate 100 mg/5 mL dry syrup was dissolved by 20 mL of water split in 2 portions. Then the drug was shaken well for at least 30 seconds at each addition of water.
  Interventions: Drug: Cefixime Trihydrate 100 mg/5 mL Dry Syrup
- Suprax® 100 mg/5 mL dry syrup (Active Comparator): Suprax® 100 mg/5 mL dry syrup was dissolved by 33 mL of water split in 2 portions. Then the drug was shaken well for at least 30 seconds at each addition of water.
  Interventions: Drug: Suprax 100 MG in 5 mL Oral Suspension

INTERVENTIONS:
Drug: Cefixime Trihydrate 100 mg/5 mL Dry Syrup — Participants received a single dose of 5 mL of cefixime dry syrup with 240 mL of water
  Arms: Cefixime trihydrate 100 mg/5 mL dry syrup
Drug: Suprax 100 MG in 5 mL Oral Suspension — Participants received a single dose of 5 mL of Suprax with 240 mL of water
  Other Names: Cefixime Trihydrate 100 mg/5 mL Dry Syrup
  Arms: Suprax® 100 mg/5 mL dry syrup

SUMMARY:
This study was conducted to investigate whether 100 mg/5 mL cefixime trihydrate dry syrup manufactured by PT. Bernofarm, Indonesia was bioequivalent to its reference product, 100 mg/5 mL Suprax® dry syrup manufactured by Odan Laboratories Ltd., Canada registered trademark of Astellas Pharma Inc., Japan.

DETAILED DESCRIPTION:
Twenty two healty subjects were given a single dose of 100 mg/5 mL cefixime trihydrate dry syrup or or 100 mg/5 mL Suprax® dry syrup with 240 mL of water. Then the blood samples for cefixime trihydrate was drawn and analyzed using HPLC. All subjects sample plasma were analyzed for pharmacokinetic evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects
2. Had read the subject information and signed informed consent documents
3. Age 18 - 55 years
4. Body mass index between 18-25 kg/m2
5. Had a normal electrocardiogram
6. Blood pressure within normal range (systolic 90-120 mmHg and diastolic 60-80 mmHg)
7. Heart rate within normal range (60-100 bpm)
8. The absence of significant disease or clinically significant abnormal laboratory values on laboratory evaluation, medical history or physical examination during screening

Exclusion Criteria:

1. those who were pregnant and/or nursing women.
2. those who had a history of contraindication or hypersensitivity to cefixime, other antibiotics or other ingredients in the drugs or a history of serious allergic reaction to any drug, significant allergic disease or allergic reaction
3. those who had a history or present medical condition which might significantly influence the pharmacokinetics of the study drug, e.g. chronic gastrointestinal disease, diarrhea, gastric surgery, renal insufficiency, hepatic dysfunction, and cardiovascular disease.
4. those who had a history or presence of any coagulation disorder or clinically significant hematology abnormalities.
5. those who were using any medication (prescription or non-prescription drug, food supplement, herbal medicine), particularly the medication known to affect the pharmacokinetics of the study drug, within one week prior to the drug administration day.
6. those who had participated in any clinical study within 3 months prior to the study (< 90 days).
7. those who had donated or lost 300 ml (or more) of blood within 3 months prior to the study.
8. those who smoked more than 10 cigarettes a day.
9. those who had a history of traveling to another city within the last 14 days
10. those with a history of direct contact with a COVID-19 positive person in the subject neighborhood
11. those with a history or presence of sore throat, fever (with temperature more than 37°C) or short of breath within the last 14 days
12. those who were positive to COVID-19
13. those who were positive to HIV, HBsAg, and HCV tests (to be kept confidential).
14. those with a history of drug or alcohol abuse within 12 months prior to screening for this study.
15. those who were unlikely to comply with the protocol, e.g uncooperative attitude, inability to return for follow-up visits, poor venous access.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2020-08-25 (Actual)

PRIMARY OUTCOMES:
Geometric Mean Ratio | 32 hours
  The ratio between test drug and reference drug
90% confidence intervals | 32 hours
  The two products are considered bioequivalent when the 90% confidence intervals of the cefixime trihydrate geometric mean ratio between test and reference product fall within the range of 80.00-125.00% for AUCt and Cmax.

SECONDARY OUTCOMES:
Pharmacokinetics parameter | 32 hours
  Maximum plasma concentration (Cmax)
Pharmacokinetics parameter | pre-dose at (0 h) and post dose at 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, 24 and 32 hours
  Area Under Curve from 0 to 32 hours (AUCt)

CONTACTS AND LOCATIONS:
Overall Officials: I Gusti Putu Bagus Diana Virgo, Study Director — PT Pharma Metric Labs, Indonesia; Arini Setiawati, Principal Investigator — PT Pharma Metric Labs, Indonesia
Locations (1):
- PT Pharma Metric Labs, Jakarta, DKI Jakarta, Indonesia

REFERENCES:
- [Background] Asiri YA, Al-Said MS, Al-Khamis KI, Niazy EM, El-Sayed YM, Al-Rashood KA, Al-Yamani MJ, Alsarra IA, Al-Balla SA. Comparative bioavailability study of cefixime (equivalent to 100 mg/5 ml) suspension (Winex vs Suprax) in healthy male volunteers. Int J Clin Pharmacol Ther. 2005 Oct;43(10):499-504. doi: 10.5414/cpp43499. PMID 16240707
- [Background] Kees F, Naber KG, Sigl G, Ungethum W, Grobecker H. Relative bioavailability of three cefixime formulations. Arzneimittelforschung. 1990 Mar;40(3):293-7. PMID 2346538
- [Background] Morais JA, Lobato Mdo R. The new European Medicines Agency guideline on the investigation of bioequivalence. Basic Clin Pharmacol Toxicol. 2010 Mar;106(3):221-5. doi: 10.1111/j.1742-7843.2009.00518.x. Epub 2010 Jan 7. PMID 20070293
- See also: Clinical Pharmacology and Biopharmaceutic Review — https://www.accessdata.fda.gov/drugsatfda_docs/nda/2013/202091Orig1s000ClinPharmR.pdf
- See also: Guideline For Good Clinical Practice — https://database.ich.org/sites/default/files/E6_R2_Addendum.pdf